CLINICAL TRIAL: NCT01472107
Title: Observational Study on Number and Outcome of Pregnancy in Childbearing Age Female Patients Treated With Chemotherapy for APL (Studies AIDA 0493, AIDA 2000)
Brief Title: Study on Number and Outcome of Pregnancy in Acute Promielocitic Leukaemia (APL) Patients Treated With Chemotherapy
Acronym: APL0511
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: APL0511
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Acute Promyelocytic Leukemia; Pregnancy
Keywords: Pregnancy; APL female patients
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The GIMEMA FOUNDATION promotes an observational (retrospective) study on number and outcome of pregnancy in childbearing age female patients treated with chemotherapy for APL. These patients were enrolled in studies AIDA0493, AIDA2000 and were in CR.

DETAILED DESCRIPTION:
Acute promielocitic leukaemia (APL) Among all the AML subtypes, APL has the distinction of being the most curable. The median age at diagnosis is 40 years, which is younger than with other AML subtypes. The fact that APL is more common in younger patients increases the likelihood that it may occur during fertile age. The introduction of ATRA and ATO has substantially modified the outcome of APL: in two successive studies 94% of patients achieved CR and the 6-yr OS rates (PETHEMA and GIMEMA) were about 80% 2,3,6.

ATRA is highly effective in APL patients, but adverse effects such as retinoic acid syndrome, arrhythmias, headache, rash, dizziness have been reported. Moreover, retinoids are known to be potent teratogens and increased rates of spontaneous abortion and major fetal abnormalities have been reported 10. Most of the cases reported suggest that ATRA is relatively safe for both mother and fetus when used in the second and third trimesters. By contrast, when it was used in the first trimester, a negative foetal outcome was reported. No data have yet been reported on the outcomes of pregnancies in young patients with APL, occurring during CCR following ATRA-including chemotherapy regimens.

APL therapy AIDA regimen: simultaneous Atra plus IDArubicin (AIDA) combination for induction treatment, followed by 3 courses of intensive chemotherapy as consolidation2.

Consolidation therapy in the AIDA-0493 trial consisted of 3 chemotherapy courses with Ara-C and idarubicin3.

Consolidation treatment in the AIDA-2000 was given according to a risk-adapted strategy as follows: patients with low-/intermediate-risk received the same 3 consolidation courses as in the AIDA-0493 but with omission of cytarabine; patients in the high-risk group received the identical 3 cycles as in the AIDA-0493.

Study rationale This is an observational (retrospective) study on number and outcome of pregnancy in childbearing age female patients treated with chemotherapy for APL. These patients were enrolled in studies studies AIDA0493, AIDA2000 and were in CR.

ELIGIBILITY:
Inclusion Criteria:

* Patients alive aged between 18 and 50 years
* Patients with unequivocal diagnosis of APL according to the FAB classification or WHO 2008 diagnostic criteria.

Female in childbearing age treated for APL, enrolled in the studies AIDA0493, AIDA2000 in CR after 2 years of maintenance with the exclusion of those randomized to observation in the AIDA2000, AIDA0493

Exclusion Criteria:

* Patients aged < 18 and > 50 years;
* Patients receiving chemotherapy;
* Concomitant psychiatric disorder that would interfere or prevent the subject from participating in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patients enrolled in studies AIDA0493, AIDA2000 in CR .
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2012-03-07 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Description of pregnancies | At 24 monhts from study entry
  The primary objective is to describe pregnancies in female patients treated with AIDA0493, AIDA2000 studies.

SECONDARY OUTCOMES:
Children's health | at 24 months from study entry
  Children's health and follow-up data
Pregnancies evolution | At 24 months from study entry
  Pregnancies evolution and outcome, children health and follow-up data according to AIDA0493 and AIDA2000 treatment strategies

CONTACTS AND LOCATIONS:
Overall Officials: Giogina SPECCHIA, Pr., Principal Investigator — UO Ematologia con trapianto- AOU Policlinico Consorziale di Bari
Locations (36):
- Italy (36):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera - Nuovo Ospedale "Torrette", Ancona
  - Unità Operativa Ematologia 1 - Università degli Studi di Bari, Bari
  - Ospedali Riuniti di Bergamo, Bergamo
  - Azienda Ospedaliera Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Sanitaria di Bolzano - Ospedale Centrale - Ematologia e Centro TMO, Bolzano
  - Sezione di Ematologia e Trapianti Spedali Civili, Brescia
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Sezione di Ematologia C.T.M.O. Istituti Ospitalieri, Cremona
  - Sez.Ematologia e Dip. scienze Biomediche Arcispedale S. Anna, Ferrara
  - Policlinico di Careggi, Università delgi studi di Firenze, Florence
  - Clinica Ematologica - DiMI - Università degli Studi di Genova, Genova
  - Divisione di Ematologia Ospedale "Santa Maria Goretti", Latina
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - Ospedale Niguarda " Ca Granda", Milan
  - U.O. Ematologia e Trapianto di MIdollo - Ist.Scientifico Ospedale San Raffaele, Milan
  - Centro Oncologico Modenese - Dipartimento di Oncoematologia, Modena
  - N. Osp. divisione di Ematologia "S.Gerardo dei Tintori", Monza
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Ospedale S. Gennaro ASL NA1, Napoli
  - Divisione di Ematologia con trapianto di midollo - A.U. Policlinico "Paolo Giaccone", Palermo
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della MIsericordia, Perugia
  - Istituto di Ematologia- Ospedale San Carlo, Potenza
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Vulture U.O. di Ematologia - Centro Oncologico Basilicata, Rionero in Vulture
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - U.O.C. di Ematolgia - A.O. " SS Annunziata" - P.O. S.G. Moscati, Taranto
  - SCDO Ematologia 2 AOU S.Giovanni Battista, Torino
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Ospedale San Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation Website — http://www.gimema.it